CLINICAL TRIAL: NCT06093932
Title: Efficacy of Songling Xuemaikang Capsules on Grade 1 Hypertension: a Randomized, Multicenter, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy of Songling Xuemaikang Capsules on Grade 1 Hypertension: a Randomized Controlled Trial
Acronym: ESCIHP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: China Academy of Chinese Medical Sciences Xiyuan Hospital Shanxi Hospital (Unknown); Suzhou Hosptial of Traditional Chinese Medicine (Unknown); China Academy of Chinese Medical Sciences Xiyuan Hospital Jining Hospital (Unknown); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023XL012-3
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Hypertension,Essential
Keywords: Songling Xuemaikang Capsules; Vascular remodeling; Grade 1 hypertension; Mild hypertension
MeSH Terms: conditions — Essential Hypertension; Vascular Remodeling | interventions — songling xuemaikang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle intervention + Songling Xuemaikang Capsules (Experimental): 1. Therapeutic Hypertensive Lifestyle Modifications, everyday, duration: 12 weeks
  2. Songling Xuemaikang Capsules, 3 capsules at a time, three times a day, duration: 12 weeks
  Interventions: Drug: Songling Xuemaikang Capsules; Behavioral: Lifestyle intervention
- Lifestyle intervention + placebo (Placebo Comparator): 1. Therapeutic Hypertensive Lifestyle Modifications, everyday, duration: 12 weeks
  2. placebo, 3 capsules at a time, three times a day, duration: 12 weeks
  Interventions: Behavioral: Lifestyle intervention; Drug: Placebo

INTERVENTIONS:
Drug: Songling Xuemaikang Capsules — 3 capsules at a time, three times a day, duration: 12 weeks
  Arms: Lifestyle intervention + Songling Xuemaikang Capsules
Behavioral: Lifestyle intervention — everyday, duration: 12 weeks
Drug: Placebo — 3 capsules at a time, three times a day, duration: 12 weeks
  Arms: Lifestyle intervention + placebo

SUMMARY:
The purpose of this study is:

1. To evaluate the efficacy of Songling Xuemaikang Capsules(SLXMKC) with grade 1 hypertension.
2. To reveal the potiential effects of SLXMKC on vascular function and structure of patients with grade 1 hypertension.
3. To explore the underlying mechanisms of the therapeutic effects of SLXMKC on the intervention of grade 1 hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35-65 years old, male or female;
* Grade 1 essential hypertension;
* Taking no antihypertensive drugs or taking antihypertensive drugs irregularly in the past ;
* Sign the informed consent;

Exclusion Criteria:

* Significant liver and kidney dysfunction, ALT and AST upper the twice of normal range, Scr≥2.0mg/dl, eGFR<60ml/(min·1. 73m2);
* Gastrointestinal diseases, which may affect drug absorption;
* Be allergic to the clinical trial medicine;
* Pregnant or breastfeeding women, men who plan to give birth within half a year;
* Combined with other serious primary diseases or malignant tumors;
* Hyperlipidemia with or without taking lipid-lowering drugs;
* Combined with left ventricular hypertrophy, ABI < 0.9, CIMT ≥ 0.9mm or atherosclerotic plaque;
* Hypertensive comorbidities (cerebrovascular disease, other cardiovascular diseases, renal disease, peripheral artery disease, retinopathy, diabetes);
* Other serious conditions in which is not fit for the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Mean 24h Systolic Blood Pressure at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)

SECONDARY OUTCOMES:
Change from Baseline in the ba-PWV at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the skin capillary density(SCD) at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Mean 24h Diastolic Blood Pressure at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Mean daytime Systolic Blood Pressure at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Mean daytime Diastolic Blood Pressure at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Mean nighttime Systolic Blood Pressure at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Mean nighttime Diastolic Blood Pressure at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Mean 24h PP at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the BP load at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Official PP at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Official SBP at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Official DBP at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Official BP Compliance Rate at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Home SBP at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Home DBP at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Proportion of patients with grade 2 or higher hypertension or target organ damage at 12 weeks | Week 12
  Proportion= Number of target patients/Total patients
Change from Baseline in the CIMT at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Hypertension Symptom Quantitative Score at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Patient Health Questionnaire-9 Quantitative Score at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)
Change from Baseline in the Generalized Anxiexy Disorde-7 Quantitative Score at 4,12 weeks | Baseline and Week 4,12
  Change=(Week 12 value- Baseline value) and (Week 4 value- Baseline value)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Xu, Prof., Study Chair — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (5):
- China (5):
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Suzhou Hosptial of Traditional Chinese Medicine, Suzhou, Jiangsu
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - China Academy of Chinese Medical Sciences Xiyuan Hospital Jining Hospital, Jining, Shandong
  - China Academy of Chinese Medical Sciences Xiyuan Hospital Shanxi Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang DY, Cheng YB, Guo QH, Shan XL, Wei FF, Lu F, Sheng CS, Huang QF, Yang CH, Li Y, Wang JG. Treatment of Masked Hypertension with a Chinese Herbal Formula: A Randomized, Placebo-Controlled Trial. Circulation. 2020 Nov 10;142(19):1821-1830. doi: 10.1161/CIRCULATIONAHA.120.046685. Epub 2020 Oct 6. PMID 33019798
- [Derived] Liu Q, Yu L, Zhang Z, Zhuang Z, Tian W, Wang A, Xu H. The effects of Songling Xuemaikang capsule on vascular remodeling of stage 1 hypertension: a multicenter, randomized placebo-controlled trial protocol. BMC Complement Med Ther. 2025 Aug 6;25(1):300. doi: 10.1186/s12906-025-05038-y. PMID 40770317